CLINICAL TRIAL: NCT06561828
Title: Developing Transcranial Neuromodulation Protocols for Learning and Decision-Making
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 10001932; 001932-DA
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-05

CONDITIONS: Normal Physiology
Keywords: TMS; Decision Making; fMRI; Learning; Behavioral Tasks

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experiment 1 (Experimental): Healthy volunteers in experiment 1
  Interventions: Device: continuous Theta Burst Stimulation (cTBS); Device: intermittent Theta Burst Stimulation (iTBS); Device: sham Theta Burst Stimulation (sham TBS)
- Experiment 2 (Experimental): Healthy volunteers in experiment 2
  Interventions: Device: continuous Theta Burst Stimulation (cTBS); Device: intermittent Theta Burst Stimulation (iTBS); Device: sham Theta Burst Stimulation (sham TBS)
- Experiment 3 (Experimental): Healthy volunteers in experiment 3
  Interventions: Device: continuous Theta Burst Stimulation (cTBS); Device: intermittent Theta Burst Stimulation (iTBS)
- Experiment 4 (Experimental): Healthy volunteers in experiment 4
  Interventions: Device: continuous Theta Burst Stimulation (cTBS)
- Experiment 5 (Experimental): Healthy volunteers in experiment 5
  Interventions: Device: continuous Theta Burst Stimulation (cTBS); Device: sham Theta Burst Stimulation (sham TBS)

INTERVENTIONS:
Device: continuous Theta Burst Stimulation (cTBS) — Continuous theta burst stimulation (three TMS pulses delivered at 50Hz with the bursts delivered at 5Hz for a total of 600 pulses per site).
Device: intermittent Theta Burst Stimulation (iTBS) — Intermittent theta burst stimulation (three TMS pulses delivered at 50Hz with the bursts delivered at 5Hz for 2 seconds followed by a break of 8 seconds for a total of 600 pulses per site).
  Arms: Experiment 1; Experiment 2; Experiment 3
Device: sham Theta Burst Stimulation (sham TBS) — iTBS or cTBS delivered with placebo side of A/P coil.
  Arms: Experiment 1; Experiment 2; Experiment 5

SUMMARY:
Background:

People with substance use disorder (SUD) often have changes in brain function that can make it difficult to control drug-seeking behavior. These changes may heighten the urge to use drugs or lessen the desire to seek nondrug-related rewards. Researchers want to know how a technique called transcranial magnetic stimulation (TMS) may cause changes in brain activity that may help people with SUD.

Objective:

To test TMS in healthy volunteers.

Eligibility:

Healthy people aged 18 to 45 years who are right-handed.

Design:

Participants can volunteer for up to 5 different experiments. Each experiment requires 2 to 8 clinic visits. Each visit will last 3 to 7 hours.

Some visits will include TMS. A coil will be placed on the participant s head. A brief electrical current will pass through the coil to create a magnetic field. Participants may feel a tapping or pulling sensation on the skin under the coil. They may feel a twitch in their face, neck, arm, or leg muscles. Participants may be asked to tense certain muscles during TMS.

Some visits will include functional magnetic resonance imaging (fMRI) scans. Participants will lie on a bed that slides into a large tube. They will perform tasks on a computer inside the tube. The fMRI will show which parts of the brain are used during each task.

Participants will perform tasks on a computer. Some tasks may be done at a desk as well as during TMS and fMRI. Participants may look at images, listen to sounds, smell odors, or taste flavored liquids. Their vital signs may be monitored and their eye movements may be tracked during tasks.

DETAILED DESCRIPTION:
Study Description:

Learning and decision-making are critical for adaptive behavior and survival. Treating maladaptive behaviors in neuropsychiatric conditions, such substance use disorder, requires knowledge about the causal neural mechanisms supporting these functions as well as ways to modulate them. The goal of the current study is to develop and validate neuromodulation protocols that target specific cognitive functions involved in learning and decision making.

Objectives:

The primary objective is to develop and validate non-invasive neuromodulation protocols that target specific cognitive functions related to learning and decision making and modulate activity in associated brain networks.

Endpoints:

The primary endpoints are to determine if the developed neuromodulation protocols reliably modulate specific cognitive functions and whether they modulate activity in the targeted brain networks.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet the following criteria:

* Willingness to comply with all study procedures and availability for the duration of the study. Consent signature will be documentation of meeting this criterion.
* Aged 18-45 years old. Justification: Many neural processes change with age, and these changes could introduce unwanted variability in the measured signals.
* In good general health based on the assessment of the MAI.
* Agreement to adhere to Lifestyle Considerations throughout study

duration. Consent signature will be documentation of meeting this criterion.

-Right-handed.

EXCLUSION CRITERIA:

Individuals who meet any of the following criteria will be excluded from participation:

* Any neurological disorder that would increase seizure risk from TMS such as stroke, brain lesions, previous neurosurgery, epilepsy, any history of seizure or fainting episode of unknown cause, frequent severe headache, or head trauma resulting in loss of consciousness, lasting over 30 minutes or with sequela lasting longer than one month. The MAI will also retain discretion to exclude based on a history of a neurological illness or trauma that may compromise safety or data integrity.
* Predisposition to seizures (e.g., first-degree family history of potentially hereditary epilepsy, etc.).
* Current use (any use in the past two weeks, daily use for more than one week within past 3 months) of any investigational drug or of any medications with psychotropic (e.g., benzodiazepines, etc.), anti or pro-convulsive action. This will be determined at the discretion of the MAI.
* Unable to undergo MRI or TMS due to certain metallic or magnetic devices or implants in the body, claustrophobia, or other reasons.
* History of noise-induced hearing loss or tinnitus.
* Recent history (within past 12 months) of learning disability, major DSM-5 psychiatric disorder including major affective disorder, ADHD, obsessive-compulsive disorder, schizophrenia, or PTSD. This will be determined at the discretion of the MAI.
* Pattern of alcohol and drug use in the past 12 months that is indicative of harmful use, loss of control over use, or physical dependence.
* Daily nicotine, alcohol, or drug use (excluding caffeine) for at least 4 continuous weeks within the past 12 months.
* Participation in any neuromodulation (e.g., TMS, tFUS, tDCS, tACS, etc.) session (excluding the current protocol) in the past two weeks.
* For tasks that involve gustatory or olfactory stimuli, food intake: History of anaphylaxis, e.g., due to severe asthma or food and non-food allergies (e.g., latex, detergents, soap, etc.). This will disqualify participants for tasks that involve chemosensory stimuli or food intake, but not from the protocol itself.
* Uncorrected impairments in visual acuity severe enough to affect task participation.
* Non-English speaking. Justification: Data integrity of some of the cognitive tasks used in this study would be compromised as they have only been validated in English. Most importantly, ongoing communication regarding safety procedures is necessary when participants are undergoing TMS and MRI procedures. The inability to effectively communicate TMS and MRI safety procedures in a language other than English could compromise the safety of non-English speaking participants.
* Pregnancy. Justification: It is unknown whether MRI and TMS pose risks to fetuses.
* Any other condition that in the judgment of the investigators is incompatible with participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2044-11-01 (Estimated); Study Completion 2044-11-02 (Estimated)

PRIMARY OUTCOMES:
Task Performance | after each intervention
  Responses on behavioral tasks

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Kahnt, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No